CLINICAL TRIAL: NCT01676246
Title: Pharmacokinetics, Metabolism and Analgesic Effects of Flupirtine After Intravenous, Single Dose and Chronic Oral Administration in Healthy Subjects Genotyped for NAT2, UGT1A1 and GSTP1
Brief Title: Pharmacokinetics, Metabolism and Analgesic Effects of Flupirtine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: AWD.pharma GmbH & Co. KG (Unknown)
Responsible Party: Principal Investigator, Prof. Werner Siegmund, Prof. Dr. W. Siegmund, MD, University Medicine Greifswald
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Flpmetab2008
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Pain; Pharmacokinetics; Flupirtine
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- flupirtine per os single dose (Active Comparator): 100 mg flupirtine per os, pharmacokinetics of flupirtine, induce delayed onset of muscle soreness (DOMS), electric pain measurement
  Interventions: Drug: 100 mg flupirtine per os; Procedure: induce delayed onset of muscle soreness (DOMS); Procedure: electric pain measurement
- flupirtine intravenous (Active Comparator): 100 mg flupirtine intravenous, pharmacokinetics of flupirtine, induce delayed onset of muscle soreness (DOMS), electric pain measurement
  Interventions: Drug: 100 mg flupirtine intravenous; Procedure: induce delayed onset of muscle soreness (DOMS); Procedure: electric pain measurement
- flupirtine per os steady state (Active Comparator): 400 mg flupirtine per os, pharmacokinetics of flupirtine, electric pain measurement
  Interventions: Drug: 400 mg flupirtine per os; Procedure: electric pain measurement

INTERVENTIONS:
Drug: 100 mg flupirtine intravenous — Administration of 100 mg flupirtine intravenous (3 mg solution intravenously, 1 vial Kadadolon® inject)
  Other Names: 1 vial Kadadolon® inject
  Arms: flupirtine intravenous
Drug: 100 mg flupirtine per os — Administration of 100 mg flupirtine per os (1 capsule Kadadolon®)
  Other Names: 1 capsule Kadadolon®
  Arms: flupirtine per os single dose
Drug: 400 mg flupirtine per os — Administration of 400 mg flupirtine (1 Kadadolon® S long retard tablet)
  Other Names: 1 Kadadolon® S long retard tablet
  Arms: flupirtine per os steady state
Procedure: induce delayed onset of muscle soreness (DOMS) — The DOMS exercise protocol consists of two sets of 50 concentric/eccentric contractions of the calf muscles of one leg with a rest of 5 min in-between. The exercise is performed 22-26 h prior to medication. For pain measurements, muscle pain is stimulated by standing on tiptoes of one leg for 30 s, which requires a constriction of the affected calf muscles. The other leg is lifted and the subjects are allowed to hold on to a table to keep their balance. The pain intensity during this stimulation is then rated by means of a 10 cm visual analogue scale (VAS). The VAS is extended from "no pain" to "intolerable pain" with a precision of 1 mm. The stimulation is repeated with the other leg. The sequence of the legs is chosen randomly.
  Arms: flupirtine intravenous; flupirtine per os single dose
Procedure: electric pain measurement — The method has been described to be sensitive to quantify analgesic opioid effects. Painful 5 Hz sine waves electrical stimuli (increase of intensity 0.2 mA/s, from 0 to 20 mA), which predominantly activate C-fibres, will be applied via two gold electrodes placed on the medial and lateral side of the distal phalangeal joint (middle finger of the left hand as default-testing site).
  During testing, subjects keep a button continuously pressed until they find the pain intolerably and interrupt the current by releasing the button. The electrical current at which this occurred is defined as pain tolerance, the target parameter of this pain model. Each value of pain tolerance is the median of five subsequent measurements obtained at an interval of 1 min.

SUMMARY:
Flupirtine is metabolized in-vitro via carbamate cleavage and N acetylation to glucuronides and mercapturic acid derivatives. The formation of reactive, toxic intermediate products may be influenced by genetic polymorphisms of the involved conjugative metabolic pathways. So the purpose of this study is to measure pharmacokinetics, metabolism and analgesic effects of flupirtine in dependence on the function of NAT2, UGT1A1 and GSTP1.

DETAILED DESCRIPTION:
Flupirtine is a centrally acting analgesic drug. Its mechanism of action differs obviously from opiates because flupirtine antagonizes the morphine-induced tail phenomenon in mice in relatively low doses. The drug exerts no relevant anesthetic activity and it has only slight inhibitory effect on prostaglandin formation in animals. As major action mechanism, activation of descending noradrenergic neuronal pathways is discussed, thereby inhibiting afferent nociceptive stimuli on spinal, subcortical and cortical brain areas. Recently has been shown, that flupirtine exhibits functional NMDA receptor antagonistic properties by selective opening the neuronal potassium channel.

The anticonvulsant drug retigabine, which chemical structure only slightly differs from flupirtine (aromatic ring instead of the pyrimidine ring), is subjected to intensive glucuronidation and N-acetylation in man. In-vitro, retigabine is a substrate of the recombinant uridine glucoronosyl transferase (UGT) 1A1, 1A3, 1A4 and 1A9. Disposition of retigabine, however, was not influenced by the frequent UGT1A1*28 polymorphism (Gilbert-Meulengracht syndrome) whereas the polymorphism of the N-acetyltransferase 2 (NAT2) resulted in significant changes in retigabine disposition.

Similar to retigabine, the carbamate group of flupirtine is hydrolyzed by carboxyl esterases. The decarbamylated product undergoes N-acetylation to form the major metabolite D13223. This acetylation is catalyzed in-vitro both by recombinant human NAT2 and NAT1. Furthermore, relatively stable quinone diimines for flupirtine and D13223 as catalyzed by peroxidases were detectable in in-vitro experiments. After repeated oral administration of flupirtine in man, quinone diimines and glutathione adducts of them in the form of mercapturic acid conjugates were detected.

Therefore, we hypothesize, that highly reactive diimine radicals may appear as intermediates which are detoxified by conjugation with glutathione via a glutathione S-transferase (GST). Diimine intermediates are known to have high cell toxicity, genotoxicity and carcinogenicity as shown for the intermediates of acetaminophen. By analogy to acetaminophen, the GSTP1 might be the isoform that is involved also in detoxification of flupirtine intermediates.

According to our hypothesis, the net appearance of toxic intermediates with diimine structure in hepatocytes is dependent on the activity of NAT1/NAT2, UGTs and GSTP1. Because NAT2, UGT1A1 and GSTP1 are highly polymorphic enzymes, the risk of flupirtine hepatotoxicity may be dependent on the genotype of the subjects that are treated with the drug.

Our clinical study was initiated to confirm, whether polymorphisms of NAT2, UGT1A1 and GSTP1 may significantly influence disposition and analgesic effect of flupirtine and whether the genetic background is of risk for the appearance of toxic intermediates and its stable terminal conjugates.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 - 45 years
* sex and genetics: male and female genotyped for NAT2, UGT1A1 and GSTP1
* ethnic origin: Whites
* body weight: 19 - 27 kg/m²
* good health as evidenced by the results of the clinical examination, ECG, and the laboratory check-up, which are judged by the clinical investigator not to differ in a clinical relevant way from the normal state
* written informed consent

Exclusion Criteria:

* existing cardiac or hematological diseases and/or pathological findings which might interfere with safety, pharmacodynamic effect and/or pharmacokinetics of the study drug
* existing or further obstructive lung disease (e.g. bronchial asthma)
* myasthenia gravis
* existing hepatic and renal diseases and/or pathological findings which might interfere with safety, pharmacodynamic effect and/or pharmacokinetics of the study drug
* existing gastrointestinal diseases and/or pathological findings which might interfere with safety, pharmacodynamic effect and/or pharmacokinetics of the study drug
* acute or chronic diseases which could affect drug absorption or metabolism
* history of any serious psychological disorder
* drug or alcohol dependence
* positive drug screening or -only in suspicious case- positive alcohol test
* smokers of 10 or more cigarettes per day
* positive screening results for HIV, HBV and HCV
* volunteers who are on a diet which could affect the pharmacokinetics of the drug (vegetarian)
* heavy tea or coffee drinkers (more than 1l per day)
* lactation and pregnancy test positive or not performed
* volunteers suspected or known not to follow instructions
* volunteers who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to as a result of their participation in the study
* volunteers liable to orthostatic dysregulation, fainting, or blackouts
* blood donation or other blood loss of more than 400 ml within the last 12 weeks prior to the start of the study
* participation in a clinical trial during the last 3 months prior to the start of the study
* less than 14 days after last acute disease
* any systemically available medication within 4 weeks prior to the intended first administration unless, because of the terminal elimination half-life, complete elimination from the body can be assumed for the drug and/or its primary metabolites (except oral contraceptives)
* repeated use of drugs during the last 4 weeks prior to the intended first administration, which can influence hepatic biotransformation (e.g. barbiturates, cimetidine, phenytoin, rifampicin)
* repeated use of drugs during the last 2 weeks prior to the intended first administration which affect absorption (e.g. laxatives, metoclopramide, loperamide, antacids, H2-receptor antagonists)
* intake of grapefruit containing food or beverages within 7 days prior to administration
* known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparation
* subjects with severe allergies or multiple drug allergies

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
bioavailability (F) | before and 0.5,1,1.5,2,2.5,3,3.5,4,5,6,8,10,12,16,24,48,72,96,120 h after administration of study medication
  ratio of the area under the concentration time curve after oral to intravenous administration of study medication
delayed onset of muscle soreness (DOMS) | before and 2, 4, 6, 8 h after study medication
  For pain measurements, muscle pain is stimulated by standing on tiptoes of one leg for 30 s, which requires a constriction of the affected calf muscles. The other leg is lifted and the subjects are allowed to hold on to a table to keep their balance. The pain intensity during this stimulation is then rated by means of a 10 cm visual analogue scale (VAS). The VAS is extended from "no pain" to "intolerable pain" with a precision of 1 mm.
electric pain threshold | before and 2, 4, 6, 8 h (and 10, 12 h on study day 8) after study medication and on study days 1,2,3,4,5,6,7
  A painful 5 Hz sine waves electrical stimuli (increase of intensity 0.2 mA/s, from 0 to 20 mA), will be applied via two gold electrodes placed on the medial and lateral side of the distal phalangeal joint (middle finger of the left hand as default-testing site). During testing, subjects keep a button continuously pressed until they find the pain intolerably and interrupt the current by releasing the button. The electrical current at which this occurred is defined as pain tolerance, the target parameter of this pain model. Each value of pain tolerance is the median of five subsequent measurements obtained at an interval of 1 min.

SECONDARY OUTCOMES:
amount of excretion (Ae) in urine | in 24 h intervals for 3 days
  urinary excretion of flupirtine, D13223 and metabolites
amount of excretion (Ae) of feces | 5 day sampling period
  fecal excretion of flupirtine, D13223 and metabolites

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Ernst-Moritz-Arndt-University Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany